CLINICAL TRIAL: NCT05173402
Title: Treating Gnathic Form of Mesial Occlusion in Early Adolescence Patients: A Clinical Trial
Brief Title: Treating Gnathic Form of Mesial Occlusion in Early Adolescence Patients
Status: Completed | Type: Observational
Sponsor: The 108 Military Central Hospital (Other Government)
Responsible Party: Principal Investigator, Le Thi Thu Hai, Dr., Associate Professor, The 108 Military Central Hospital
Other Study IDs: Le Thi Thu Hai
Record Dates: First submitted 2021-12-14; First posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Gnathic (Skeletal) Mesial Occlusion
Keywords: early adolescence; orthodontic practice; orthodontic treatment
MeSH Terms: interventions — Masks

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The experimental group: The experimental group included 26 patients - orthopedic treatment was performed using the dentoalveolar compensation method with permanent apparatus with a palatal expanding screw.
  Interventions: Device: dentoalveolar compensation method
- The comparison group: The comparison group included 20 patients - orthopedic treatment was performed using a face mask.
  Interventions: Device: face mask

INTERVENTIONS:
Device: dentoalveolar compensation method — orthopedic treatment was performed using the dentoalveolar compensation method with permanent apparatus with a palatal expanding screw
  Groups: The experimental group
Device: face mask — orthopedic treatment was performed using a face mask.
  Groups: The comparison group

SUMMARY:
The primary purpose of this study was to evaluate the immediate and previous results of the effectiveness of non-surgical orthopedic treatment in children aged 12-14 years with gnathic forms of mesial occlusion by the method of dentoalveolar compensation using a permanent apparatus with a palatal expanding screw.

ELIGIBILITY:
Inclusion Criteria:

patients with a gnathic (skeletal) mesial occlusion patients age 12-14 years patients who underwent orthopedic treatment

Exclusion Criteria:

change of residence severe form of gnathic mesial occlusion congenital anomalies of the dento-maxillo-facial area

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: To evaluate the early and late results of the non-surgical orthopedic treatment efficiency in 12-14 years old children with the gnathic forms of mesial occlusion by the dentoalveolar compensation utilizing a permanent device with a palatal expanding screw.
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2014-09-05 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
dentoalveolar compensation method | 2014-2020
  orthopedic treatment was performed using the dentoalveolar compensation method with permanent apparatus with a palatal expanding screw
face mask | 2014-2020
  orthopedic treatment was performed using a face mask

IPD SHARING:
Plan to Share IPD: No
The study was anonymous. No personal data will be revealed